CLINICAL TRIAL: NCT02402322
Title: Internet-based Self-help Treatment for Panic Disorder: A Randomised Controlled Trial of Two Ways of Administrating the Complementary Psychological Support (Scheduled vs. Non-scheduled)
Brief Title: Internet-based Self-help Treatment for Panic Disorder: Two Ways of Complementary Psychological Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Pablo Oromendia, PhD Candidate, Universitat Autonoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTCCAP
Record Dates: First submitted 2015-03-20; First posted 2015-03-30 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-10

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-scheduled support (Active Comparator): Participants received an Web-based cognitive behavioral treatment for Panic Disorder with the support of a therapist via phone when they required it.
  Interventions: Behavioral: Non-scheduled support
- Scheduled support (Experimental): Participants received an Web-based cognitive behavioral treatment for Panic Disorder with the support of a therapist via phone weekly.
  Interventions: Behavioral: Scheduled support
- Waiting list (No Intervention): Participants in a waiting list.

INTERVENTIONS:
Behavioral: Scheduled support — Participants followed the online self-help program based on cognitive behavioral therapy for 8 weeks. They had the support of a therapist via phone weekly.
  Arms: Scheduled support
Behavioral: Non-scheduled support — Participants followed the online self-help program based on cognitive behavioral therapy for 8 weeks. They had the support of a therapist via phone when they required it.
  Arms: Non-scheduled support

SUMMARY:
The aim of this study was to compare two ways of administrating the complementary psychological support (scheduled vs. non-scheduled) in an online self-help program for panic disorder. In order to do so, the investigators studied: a) If there were differences in the intensity and frequency of the symptoms of panic disorder. b) If there were differences in the therapeutic adherence between the subjects receiving both kinds of complementary support. c) If the more time spent by a psychologist in therapeutic interventions produced the best results of therapeutic adherence / symptom improvement.

Seventy seven subjects followed the online self-help program for 8 weeks; 27 subjects had the support of a therapist via phone when they required it, 25 subjects had the support of a therapist weekly and 25 subjects were in the waiting list as a control group.

DETAILED DESCRIPTION:
The aim of this study was to compare two ways of administrating the complementary psychological support (scheduled vs. non-scheduled) in an online self-help program for panic disorder. In order to do so, the investigators studied: a) If there were differences in the intensity and frequency of the symptoms of panic disorder. b) If there were differences in the therapeutic adherence between the subjects receiving both kinds of complementary support. c) If the more time spent by a psychologist in therapeutic interventions produced the best results of therapeutic adherence / symptom improvement.

Treatment program

Internet-based self-help program for anxiety disorders "FREE OF ANXIETY" was developed, based on cognitive behavioral therapy. The program is presented as an interactive course, which is divided into eight weekly modules.A number of therapeutic components are used: psychological education (modules 1-8), behavioral analysis (safety and avoidance behavior) (module 2), in vivo and interoceptive exposure (modules 2-8), relaxation training and diaphragmatic breathing (modules 1-4), cognitive restructuring (modules 4-5), mindfulness (Module 6) communication training (module 7), problem solving Module 8). The program also includes a messaging system between therapists and subjects.

Participants and Procedure

The participants were recruited using a google banner linked to searches about anxiety disorders. The individuals were redirected to a Web page which contained information about anxiety disorders and the aims of the study. Suicide risk (score of 3 in the 15th item of the Web Screening Questionnaire) was established as an exclusion criterion. The study was approved by the ethics committee of the Autonomous University of Barcelona.

Applicants completed the informed consent, the demographic questionnaire and a screening questionnaire online. One week later a psychologist who had been trained to apply the MINI International Neuropsychiatric Interview (Sheehan, Lecrubier, Harnett-Sheehan, Janavs,Weiller, Bonora, et al., 1997) assessed the presence of a current psychiatric diagnosis. Participants with Panic Disorder completed a battery of self-reported measures in order to assess panic disorder, anxiety, and depression symptoms.

After clinical evaluation, the participants were divided into three groups by a true random-number service.

The data collected were anonymized and coded

Seventy seven subjects followed the online self-help program for 8 weeks; 27 subjects had the support of a therapist via phone when they required it, 25 subjects had the support of a therapist weekly and 25 subjects were in the waiting list as a control group.

Participants completed self-reported measures at the end of the treatment, and six months later.

Statistical analyses

The investigators studied differences between participants with and without Panic Disorder regarding their gender and age, using Chi-square test and Student t-test.

The participants' pretreatment and posttreatment measures were analyzed with analysis of variance (ANOVA) with repeated measures. These were followed by t tests with Bonferroni-corrected p values. Effect sizes were calculated both within and between groups, and all calculations were based on the pooled standard deviation, Cohen's d.

All analyses were conducted using SPSS version 22 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic Statistical Manual criteria for panic disorder.
* Have suffered from panic disorder at least one year.
* Suffer from panic disorder as primary pathology.
* If the participant was taking medication for panic disorder / agoraphobia, the dose should be stable three months before the start of the program.

Exclusion Criteria:

* Obtain a score of 26 or more on the Beck Depression Inventory II
* Suffer from another psychiatric illness that requires immediate attention.
* Risk of suicide, indicated by a score of 3 on the screening questionnaire.
* Being or having been in cognitive behavioral therapy .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Molinuevo, PhD, Study Director — Department of Psychiatry and Forensic Medicine, Institute of Neurosciences, School of Medicine, Universitat Autònoma de Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements on the Internet and were redirected to a website containing information about the study. Individuals interested in taking part in the study completed a screening questionnaire and provided demographic data. Participants were recruited between August, 2013 and February 2014.
Pre-assignment Details: Individuals were evaluated thoroughly using the MINI International Neuropsychiatric Interview.
  One hundred and twenty-five individuals were assessed and 48 were excluded from the trial because they suffered from another disorder (n=34), their medication was not stable (n = 13), or they had received Cognitive Behavioral Therapy (n = 1).
Period: Pretreatment
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Started | 27 | 25 | 25
Posttreatment Measures | 24 | 24 | 24
Completed | 24 | 24 | 24
Not Completed | 3 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 1
Period: Follow-up
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Started | 24 | 24 | 24 (These individuals were not evaluated at this follow-up as they started an alternative treatment.)
Completed | 18 | 21 | 0
Not Completed | 6 | 3 | 24
Not completed — Withdrawal by Subject | 6 | 3 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List | Total
Number analyzed (Participants) | 27 | 25 | 25 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (8.5) | 38.2 (7.8) | 44.6 (10.3) | 40.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 15 | 53
  Male | 8 | 6 | 10 | 24
Region of Enrollment [Number; unit: participants]
  Spain | 27 | 25 | 25 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Score in the Panic Disorder Severity Scale at 8 Weeks and 6 Months.
Description: Panic Disorder Severity Scale Self-Report (PDSS-SR). This 7-item scale assesses the severity of PD through questions about the frequency of panic attacks, associated distress, anticipatory anxiety, agoraphobic and interoceptive avoidance, and social and work impairment. Score range: 0-28. Scores up to 10 correspond with ''mild,'' those between 11 and 15 with ''moderate,'' and those at or above 16 with ''severe'' panic disorder.
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-28)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-28)
  Base line | 15.29 (4.21) | 15.75 (4.52) | 13.08 (3.81)
  8 weeks | 10.42 (3.14) | 7.21 (2.16) | 13.13 (4.5)
  Six months | 10.21 (2.57) | 8.33 (2.61) | 13.13 (4.5)
Statistical Analysis 1: Comparison: Non-scheduled Support vs Scheduled Support vs Waiting List; The participants' pre- and posttreatment scores were studied with repeated measures ANOVA. Within- and between-group effect sizes were calculated using the pooled standard deviation, Cohen's d; Test type: Non-Inferiority or Equivalence — In the preliminary analysis, we studied the possible group differences in demographic data and pretreatment measures with chi-square tests and analysis of variance (ANOVA); p = 0.05, ANOVA

2. Primary Outcome: Change From Baseline Score in the Anxiety Sensitivity Index-3 at 8 Weeks and 6 Months.
Description: This 18-item scale evaluates sensitivity to anxiety symptoms on 3 dimensions: physical, cognitive, and social.There are 3 subscales, physical, cognitive, and social. For both the subscales (which range from 0 to 24) and the total scale (which range from 0 to 72), higher scores correspond to greater anxiety sensitivity.
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-72)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-72)
  Base line | 31.04 (10.13) | 29.00 (9.7) | 26.83 (11.56)
  8 weeks | 21.54 (10.07) | 14.75 (7.71) | 28.08 (11.94)
  6 months | 22.17 (9.86) | 16.13 (9.82) | 28.08 (11.94)

3. Secondary Outcome: Change From Baseline Score in the Beck Anxiety Inventory at 8 Weeks and 6 Months.
Description: Beck Anxiety Inventory (BAI), Spanish adaptation . This 21-item self-reported instrument evaluates the cognitive and physical symptoms of anxiety. Score range:0- 63, with 3 levels of severity 0-21 mild anxiety, 22-35 moderate anxiety and 36-63 severe anxiety.
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-63)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-63)
  Base line | 34.92 (8.6) | 34.29 (10.97) | 30.63 (9.53)
  8 weeks | 24.04 (8.84) | 16.50 (8.99) | 31.71 (10.26)
  6 months | 24.33 (9.51) | 17.75 (8.72) | 31.71 (10.26)

4. Secondary Outcome: Change From Baseline Score in the Beck Depression Inventory at 8 Weeks and 6 Months.
Description: Beck Depression Inventory-II (BDI-II), Spanish adaptation (38, 39). This 21-item self-reported instrument evaluates symptoms of depression. Score range:0- 63, with 3 levels of severity, 10-18 mild depression, 19-29 moderate depression and >30 severe depression.
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-63)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-63)
  Base line | 18.00 (5.26) | 19.46 (5.11) | 19.75 (4.77)
  8 weeks | 11.92 (6.02) | 10.71 (5.56) | 19.58 (6.71)
  6 months | 11.63 (5.33) | 10.21 (4.79) | 19.58 (6.71)

5. Secondary Outcome: Change From Baseline Score in the Sheehan Disability Inventory (Work Subscale) at 8 Weeks and 6 Months.
Description: This 5-item instrument assesses functional impairment at work, and in social and family life. There are 5 subscales: work, social life, family life, stress, social support. The first three subscales range from 0 to 10, with higher scores indicating greater disability. The fourth subscale (stress) range from 0 to 10, with higher scores indicating greater stress perceived. The fifth subscale (Social Support Subscale) ranges from 0 to 100, with higher scores indicating greater social support perceived.There is not a total score.
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-10)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-10)
  Base line | 6.33 (2.53) | 5.88 (2.61) | 5.67 (3.29)
  8 weeks | 4.42 (2.55) | 2.96 (2.42) | 5.79 (3.09)
  6 months | 4.21 (2.12) | 3.08 (2.33) | 5.79 (3.09)

6. Secondary Outcome: Change From Baseline Score in the Sheehan Disability Inventory (Social Life Subscale) at 8 Weeks and 6 Months.
Description: as for outcome 5
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-10)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-10)
  Base line | 6.25 (2.36) | 6.83 (2.27) | 5.46 (3.0)
  8 weeks | 4.54 (2.37) | 3.75 (2.48) | 5.46 (3.06)
  6 months | 4.33 (2.37) | 3.21 (2.16) | 5.46 (3.06)

7. Secondary Outcome: Change From Baseline Score in the Sheehan Disability Inventory (Family Subscale) at 8 Weeks and 6 Months.
Description: as for outcome 5
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-10)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-10)
  Base line | 4.96 (2.75) | 4.88 (2.55) | 4.58 (2.99)
  8 weeks | 3.58 (2.33) | 2.88 (2.47) | 5.21 (3.12)
  6 months | 3.46 (2.51) | 2.54 (2.57) | 5.21 (3.12)

8. Secondary Outcome: Change From Baseline Score in the Sheehan Disability Inventory (Stress Subscale) at 8 Weeks and 6 Months.
Description: as for outcome 5
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-10)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-10)
  Base line | 7.42 (1.61) | 7.38 (2.37) | 7.17 (2.29)
  8 weeks | 5.04 (2.07) | 4.63 (2.88) | 6.96 (2.86)
  6 months | 4.92 (2.10) | 3.79 (2.50) | 6.96 (2.86)

9. Secondary Outcome: Change From Baseline Score in the Sheehan Disability Inventory (Social Support Subscale) at 8 Weeks and 6 Months.
Description: as for outcome 5
Time Frame: Baseline, 8 weeks, 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale (range= 0-100)
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Number analyzed (Participants) | 24 | 24 | 24
units on a scale (range= 0-100)
  Base line | 58.75 (31.80) | 60.00 (30.78) | 49.58 (35.19)
  8 weeks | 62.92 (28.51) | 72.50 (24.53) | 62.92 (27.73)
  6 months | 68.33 (20.57) | 70.00 (22.26) | 62.92 (27.73)

ADVERSE EVENTS:
Time Frame: 8 months
Description: A weekly questionnaire regarding anxiety symptoms was administered.
Arm/Group | Non-scheduled Support | Scheduled Support | Waiting List
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No